CLINICAL TRIAL: NCT03966703
Title: Masticatory Efficiency in Implant-fixed Complete Dentures Compared to the Conventional Dentures: a Randomized Clinical Trial by Color Mixing Analysis Test.
Brief Title: Masticatory Efficiency in Implant-fixed Complete Dentures Compared to the Conventional Dentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, Elie Jasser, Master student in aesthetic and prosthetic dentistry. Principal investigator, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: USJ -2017-65
Record Dates: First submitted 2019-05-22; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Mastication
Keywords: complete denture; implant-fixed denture; masticatory efficiency; mixing ability test

STUDY DESIGN:
Intervention Model Description: 10 patients from each group
Who Masked: Participant
Masking Description: patients are computer sorted in each group. samples were anonymous tagged by numbers and not by patient name
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional denture (Experimental): 10 patients chewed a 2 color gum for 5 cycles 10, 15 and 20.each sample is retrieved weighted and scanned
  Interventions: Behavioral: mixing analysing test
- implant fixed denture (Experimental): 10 patients chewed a 2 color gum for 5 cycles 10, 15 and 20.each sample is retrieved weighted and scanned
  Interventions: Behavioral: mixing analysing test

INTERVENTIONS:
Behavioral: mixing analysing test — The chewed gum is retrieved scanned and weighted to quantify masticatory efficiency
  Other Names: gum weight; hubba bubba

SUMMARY:
Purpose of this study is to compare the masticatory efficiency 'All on four' to 'Complete dentures on a class I ridge' with a color mixing analyzing test. Ten Patients with fixed complete dentures on implants and other ten patients with complete denture on a class I ridge (Atwood) had chewed a bicolor chewing gum (Hubba Bubba ®) for different number of cycles(5-10-15-20). The chewed gum is retrieved scanned and weighted to quantify masticatory efficiency

ELIGIBILITY:
Inclusion Criteria:

* good general health, good intraoral conditions, and dentures in satisfactory conditions over edentulous high ridge Atwood's Class I. The minimum time of complete denture use ranged from 3 to 6 months. no temporomandibular dysfunction

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
color analysis mixing test | from 5 up to 20 second
  a two color chewing gum is chewed for a specific number of cycles, gum is scanned and color mixing is analysed by a software called View Gum

SECONDARY OUTCOMES:
weight reduction | from 5 up to 20 second
  gum is weighted before each chewing cycle than dried and weighted after chewing.weight reduction is the secondary outcome for mastication efficiency analyzing

CONTACTS AND LOCATIONS:
Overall Officials: Elie Jasser, DSD, Principal Investigator — Master student in aesthetic and prosthetic dentistry
Locations (1):
- Saint Joseph University, Beirut, Lebanon